CLINICAL TRIAL: NCT03846609
Title: A Randomized Controlled Study Evaluating the Performance of a Double Balloon Interventional Platform (DiLumen) for Facilitating Complex Colonic ESD
Brief Title: Evaluation of a Double Balloon Interventional Platform (DiLumen) for Complex Colonic ESD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mercy Medical Center (Other)
Responsible Party: Principal Investigator, Sergey Kantsevoy, M.D., Ph.D., Director of Therapeutic Endoscopy, Mercy Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1368768-2
Record Dates: First submitted 2019-02-12; First posted 2019-02-19 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Colonic Polyp
Keywords: Endoscopic Submucosal Dissection
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Intervention Model Description: The patients will be assigned into study group [procedure performed with use of double balloon interventional platform (DiLumen)] or control group [procedure done without the use of double balloon interventional platform (DiLumen)]
Who Masked: Participant
Masking Description: The patients will be randomly assigned to study or control group. The patients will not know their assignment until completion of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- double balloon platform (Experimental): Device: double balloon interventional platform (DiLumen)
  Interventions: Device: double balloon interventional platform (DiLumen)
- no double balloon platform (Active Comparator): Device: no double balloon interventional platform (DiLumen)
  Interventions: Device: no double balloon interventional platform (DiLumen)

INTERVENTIONS:
Device: double balloon interventional platform (DiLumen) — double balloon interventional platform (DiLumen) is used for removal of colonic polyp
  Arms: double balloon platform
Device: no double balloon interventional platform (DiLumen) — double balloon interventional platform (DiLumen) is not used for removal of colonic polyp
  Arms: no double balloon platform

SUMMARY:
The purpose of this randomized study is to compare ESD procedural time and cost facilitated with a dual balloon accessory device versus ESD procedures performed without the accessory device. Study is designed to detect if the double balloon interventional platform helps to perform removal of benign complex colonic lesions safer and in more efficient way.

DETAILED DESCRIPTION:
This is a prospective, post-market, randomized clinical trial comparing colonic ESD procedures utilizing the DiLumen™ Endolumenal Interventional Platform to colonic ESD procedures that are performed without use the DiLumen™ device.

The study participants will be randomly assigned to study group and control group The treatment group will consist of up to 100 subjects treated with the DiLumen™ device. The control group will consist of up to 100 subjects treated without DiLumen™ device. Assessments will include procedure timepoints, anesthesia use, polyp location and classification, over-all cost assessment, and general complications.

The primary outcome will be analyzed using parametric statistics to compare the means of the study and control groups. P-values and confidence intervals will be reported. Descriptive and summary statistics will also be employed. Secondary outcomes will be summarized with descriptive statistics.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women 18-85 years of age.
2. Have ability to understand the requirements of the study and provide written informed consent
3. Suspected complex adenomatous polyps in the large intestine defined as sessile or polypoid lesions 2 cm and larger in size.
4. No medical contraindication to endoscopic submucosal dissection (ESD).

Exclusion Criteria:

1. Contraindication to colonoscopy, such as active colitis, diverticulitis, perforation, or stricture.
2. History of open or laparoscopic colorectal surgery.
3. History of Inflammatory Bowel Disease (IBD).
4. Any medical or surgical condition that would preclude the endoscopic removal of the polyp.
5. Anatomy or other factors that prohibit safe access to the large intestine such as previous radiation therapy to the affected area, known colonic strictures, extensive colonic diverticuli, etc.
6. History of AIDS, HIV, or active hepatitis.
7. History of mental illness, including psychological or neurological conditions (addiction to substances such as alcohol. e.g.) that in the investigator's opinion would pre-empt their ability or willingness to participate in the study.
8. Patients who are pregnant or lactating.
9. Currently involved in another investigational product for similar purposes.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2019-02-19 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-12-10 (Actual)

PRIMARY OUTCOMES:
Total case time | 3-month
  Time from the beginning of procedure until the end of the entire procedure Iin minutes)

SECONDARY OUTCOMES:
Navigation time | 3-month
  Time from endoscope insertion into patient's rectum till colonic lesion is reached (in minutes)
Dissection time | 3-month
  Time from the start of lesion removal till the lesion removal is completed (in minutes)
Length of Hospital Stay | 3-month
  Days of admission to the hospital post procedure till the patient is discharged from the hospital (in days)
Cost of service | 3-month
  Total financial cost (in USA dollars) of the medical care received pertaining to the procedure and related follow-up
30-day readmittance rate | 30-day
  Number of patients readmitted to the hospital during first 30 days post colonoscopy
Patient satisfaction survey | 3-month
  Patients are given three statements regarding their procedures for which they answer if they agree or disagree with the statement.
Histologic pathology summary | 3-month
  The final pathological determination of the excised specimen, as determined by pathological examination
Rate of complications | 3-month
  Adverse effects that occur during the study

CONTACTS AND LOCATIONS:
Overall Officials: Sergey V Kantsevoy, MD, PhD, Principal Investigator — Director of The Therapeutic Endoscopy Mercy Medical Center
Locations (1):
- Mercy Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Study records should be stored in a secure area to limit access to study personnel and maintain confidentiality of the records.

REFERENCES:
- [Derived] Kantsevoy SV, Palmer A, Hockett D, Vilches A. Prospective, randomized controlled study evaluating a double-balloon interventional endoscopic platform for colorectal endoscopic submucosal dissection (with video). Gastrointest Endosc. 2025 Jan;101(1):149-157. doi: 10.1016/j.gie.2024.07.001. Epub 2024 Jul 5. PMID 38971202